CLINICAL TRIAL: NCT04004910
Title: A Multicenter, Open-Label, Three-Part Study to Evaluate the Safety and Effectiveness of Immunopheresis With Immunicom's LW-02 Device in Removal of Soluble Tumor Necrosis Factor Receptors (sTNF-Rs) as Well as Clinical Efficacy in Treatment of Patients With Advanced, Refractory Breast Cancer (BC) Alone, or in Combination With Low Dose Chemotherapy Versus Low Dose Chemotherapy.
Brief Title: A Study Comparing Immunopheresis® Alone or In Combination With Chemotherapy Versus Chemotherapy Alone in Treatment of Advanced Breast Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunicom Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP7-005
Record Dates: First submitted 2019-06-24; First posted 2019-07-02 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Advanced Breast Cancer
Keywords: Advanced Breast Cancer; Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; Antineoplastic Agents

STUDY DESIGN:
Intervention Model Description: A Multicenter, Open-Label, Three-Part Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immunopheresis® - Arm 1 (Experimental): All patients will receive up to 16 weeks of initial treatment as per study arm assignment, which will include up to 48 LW-02 column-based Immunopheresis® treatments over a 4-month period (up to 3 procedures per week) though treatment can be extended based on certain protocol-specfied conditions. Each patient assigned to the treatment with LW-02 column-based Immunopheresis® will require central vascular access for the procedure. This part is alrady completed.
  Interventions: Other: Plasma soluble TNF receptor pulldown
- Immunopheresis® combined with low dose chemotherapy - Arm 2 (Experimental): All patients will receive up to 16 weeks of treatment as per study arm assignment, which will include up to 48 LW-02 column-based Immunopheresis® treatments over a 4-month period (up to 3 procedures per week) though treatment can be extended based on certain protocol-specfied conditions. Each patient will require central vascular access for the procedure. Patients also will receive a low dose chemotherapy regimen administered iv or oraly. Patients treated with combination will be administered their chemotherapy following the first LW-02 column-based Immunopheresis® procedure of each week starting from week 2, assuming first week of study treatment serves as a run-in period confirming good tolerance of Immunopheresis® alone.
  Interventions: Other: Plasma soluble TNF receptor pulldown + chemotherapy
- Chemotherapy - Arm 3 (Active Comparator): Patients who are assigned chemotherapy arm of the study will be treated with low dose chemotherapy alone. The chemotherapy will be administered intravenously or oraly depending on the regimen used.
  Interventions: Drug: Chemotherapy Drugs, Cancer

INTERVENTIONS:
Other: Plasma soluble TNF receptor pulldown — The Immunoadsorption affinity column, the LW-02 column, uses a proprietary human recombinant protein, single chain TNF-α ligand, covalently linked to a bead resin, that both enhances the capture efficiency of sTNF-Rs while avoiding complications from column leaching. Reduced sTNF-R plasma levels may lead to objective tumor responses.
  Arms: Immunopheresis® - Arm 1
Other: Plasma soluble TNF receptor pulldown + chemotherapy — The Immunoadsorption affinity column, the LW-02 column, uses a proprietary human recombinant protein, single chain TNF-α ligand, covalently linked to a bead resin, that both enhances the capture efficiency of sTNF-Rs while avoiding complications from column leaching. Reduced sTNF-R plasma levels may lead to objective tumor responses.
  In combined treatment arm the Immunopheresis® procedure is combined with low dose chemotherapy to potentially enhancing the latter's cytotoxic effect.
  Arms: Immunopheresis® combined with low dose chemotherapy - Arm 2
Drug: Chemotherapy Drugs, Cancer — Low dose chemotherapy will be provided to patient either IV or oraly depending on the regimen used.
  Arms: Chemotherapy - Arm 3

SUMMARY:
This is a multicenter, open-label, Phase 1/ 2 study to evaluate the short-term and longer-term safety, tolerability, and effectiveness of Immunopheresis® with the LW-02 column in removal of Soluble Tumor Necrosis Factor Receptors (sTNF-Rs) from plasma of patients with advanced, refractory Breast Cancer (BC) and for disease control when employed as monotherapy, or in combination with a low dose chemotherapy. A low dose chemotherapy will serve as control.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase 1/ 2 study to evaluate the short-term and longer-term safety, tolerability, and effectiveness of Immunopheresis® with the LW-02 column in removal of sTNF-Rs from plasma of patients with advanced, refractory BC and for disease control when employed as monotherapy, or in combination with a low dose chemotherapy. A low dose chemotherapy will serve as control.

Part A (n=10 evaluable patients): Overall safety, tolerability, and sTNF-R-removal effectiveness of LW-02 device-based immunopheresis monotherapy conducted 3 times per week for 4 weeks in patients with advanced TNBC. This part is already completed.

Part B/Part B Extension (n = up to 30 evaluable patients): Overall safety, tolerability, and sTNF-Rs-removal effectiveness of LW-02 device-based Immunopheresis® 3 times per week for up to 16 weeks combined with low dose chemotherapy in patients with advanced refractory BC..

Part C (3 treatment arms; n=50 patients per treatment arm): Randomized comparison of overall safety, tolerability, and clinical efficacy effectiveness of (i) Immunopheresis® monotherapy with the LW-02 column 3 times per week for 16 weeks, (ii) or Immunopheresis® in combination with low dose chemotherapy, and (iii) plain low dose chemotherapy.

Safety Endpoints

1. Safety and tolerability - incidence of Adverse Device Effects (ADEs), Serious Adverse Device Effects (SADEs) and Unanticipated Serious Adverse Device Effects (USADEs) related to immunopheresis procedure as well as Adverse Events (AE) and Serious Adverse Events (SAEs).
2. Safety endpoints of special interest - incidence of tumor lysis syndrome, and systemic inflammatory response syndrome.
3. Patient-Reported Outcomes to evaluate health status and Quality of Life (QoL) instruments for patients with BC:

   * Eastern Cooperative Oncology Group (ECOG) status
   * EQ-5D-5L index-based scale
   * EORTC: QLQ-BR23 (breast), and QLQ-C30 (general cancer questionnaire)
   * 6-minute walk test and BORG dyspnea, fatigue scale and hand grip test
   * Nutritional status will be assessed with PG-SGA scale and via laboratory assessments of changes in serum albumin and CRP

Efficacy Endpoints

1. Column efficiency and effectiveness in removal of sTNF-Rs from patient plasma without clinically-meaningful leaching of capture ligand (SC-TNF-α) - change in sTNF-R and TNF-α plasma levels from initiation to the end of each Immunopheresis® procedure, including pre- and post-column measurements, between each treatment, and from baseline to end of a treatment cycle (4 weeks - Part A and B/B-extension, or 16 weeks - Part C).
2. Clinical endpoints - response in tumor burden - progression-free survival (PFS), disease control rate (DCR), objective response rate (ORR), clinical benefit rate (CBR), duration of response (DOR), duration of clinical benefit (DOCB), time-to-progression (TTP) and overall survival (OS). Serial evaluation of tumor burden/tumor growth is assessed according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1).

ELIGIBILITY:
This study will enroll approximately 170 patients with measurable advanced, refractory breast cancer [BC] (incurable stage III and stage IV) histologically confirmed and with ECOG performance status of 0, 1 and 2 who:

* are primarily diagnosed with advanced disease or are diagnosed with incurable recurrent disease and who have progressed at least 2 standard systemic treatments (with different treatment regimens)
* have not refused standard-of-care therapies

  * Prior radiation therapy is allowed, provided that the patient has recovered from any toxic effects thereof; radiotherapy will not be counted as the treatment line
  * Chemotherapy regimens will be counted based on interval disease progression, and not on the number of agents or the number of switches in agents
  * Patients with ER+ tumors must have failed at least one line of palliative endocrine treatment .
  * Patients with HER2+ tumors must have failed at least two lines of palliative anti-HER2 therapy

Inclusion Criteria:

1. Signed Informed Consent Form
2. Age ≥ 18 years female
3. Able to comply with the study protocol in the investigator's judgment
4. Histologically confirmed diagnosis of BC
5. Inoperable locally-advanced or metastatic disease
6. Must be able to provide archival pathological material from primary or metastatic site (formalin-fixed paraffin embedded [FPPE] tissue block) for central BC confirmation and verification of BC subtype and tmTNF expression
7. Weight ≥ 35 kg
8. Life expectancy of at least 3 months with malignancy; expected to live for one year without malignancy.
9. Adequate organ function:

   1. Hemoglobin ≥ 9.5g/dL (may be achieved with transfusion support)
   2. Absolute Granulocyte Count (ANC) ≥1.5 × 109/L (without granulocyte colony- stimulating factor support within 2 weeks prior to the first study treatment)
   3. Platelets (PTL) ≥ 100 × 109/L
   4. AST/ALT ≤2.5× ULN (patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN; patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 ×ULN)
   5. Serum creatinine (S-Cr) ≤ 1.5
   6. Albumin ≥ LLN
   7. Bilirubin ≤ 1.5 ULN
   8. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. This applies only to patients who are not receiving therapeutic anticoagulation agents.
   9. Patients receiving therapeutic anticoagulation agents must be on a stable dose
   10. Calcium level within normal ranges.
10. The last dose of prior systemic anticancer therapy must have been administered ≥ 7 days prior to study treatment initiation
11. Measurable disease, as defined by RECIST v1.1
12. ECOG performance status 0, 1 or 2.
13. Patients with asymptomatic CNS metastases (treated or untreated), as determined by CT or MRI evaluation during screening and prior radiographic evaluation, are eligible.
14. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use double barrier contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of chemotherapy.
15. Patients must have recovered (i.e., improvement to Grade 1 or better) from all acute toxicities from previous therapy, excluding alopecia. If a patient was previously treated with taxanes, the patient must have recovered from any adverse effects or remain at an acceptable level for patient (i.e. peripheral neuropathy).

Exclusion Criteria:

1. Symptomatic CNS metastases
2. Subjects with brain metastases at screening must have clinically controlled neurologic symptoms and have received previous adequate treatment, defined as surgical excision and/or radiation therapy with stable neurologic function and no evidence of CNS disease progression as determined by comparing a computed tomography (CT) scan or magnetic resonance imaging (MRI) scan performed during screening to a prior scan performed at least 4 weeks earlier and provided that the subject is asymptomatic, has no evidence of cavitation or hemorrhage, and does not require corticosteroids;
3. Leptomeningeal disease
4. Uncontrolled pericardial effusion or ascites requiring recurrent drainage procedures
5. Pregnant or lactating or intending to become pregnant during the study - women who are not postmenopausal (postmenopausal defined as ≥ 12 months of non-drug-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 2 weeks prior to initiation of study treatment
6. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome)
7. Significant cardiovascular disease, such as New York Heart Association cardiac disease ≥ Class III, myocardial infarction within 3 months, unstable arrhythmias, or unstable angina
8. Patients with known coronary artery disease or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
9. Patient with known persistent, uncontrolled hypotension
10. Significant renal disorder requiring dialysis or indication for renal transplant
11. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to study treatment initiation
12. Major surgical procedure within 4 weeks prior to study treatment initiation or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
13. Fever, or any active immunosuppressive systemic infection including history of human immunodeficiency virus (HIV) infection
14. Other serious diseases (e.g., life expectancy less than 3 months) including active second malignancy except for basal cell carcinoma or cervical carcinoma in situ
15. Active infection
16. Patients in whom vascular access is not considered achievable
17. Use of any standard high dose or low dose chemotherapy or immunosuppressive therapies and or standard radiation therapy concurrently as well anticipated need for any of the former during the study
18. Body mass index (BMI) ≥ 35 kg/m2
19. Any condition that the patient's physician determines to be detrimental to the patient participating in this study; including any clinically important deviations from normal clinical laboratory values or concurrent medical events.
20. Inability to understand the local language for use of the patient QOL instruments (EQ-5D-5L and others).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Soluble Tumor Necrosis Factor Receptor (sTNFR) concentrations in plasma (picogram per mL) | 16 weeks
  Column efficiency and effectiveness in removal of sTNF-Rs from patient plasma without clinically-meaningful leaching of capture ligand (SC-TNF-α) - change in sTNF-R and TNF-α plasma levels from initiation to the end of each immunopheresis procedure, including pre- and post-column measurements, between each treatment, and from baseline to end of a treatment cycle (4 weeks - Part A and B, or 16 weeks - Part C).
Safety and Tolerability Assessment | 16 weeks
  Safety and tolerability assessment based on adverse event / serious adverse event (AE / SAE) and adverse device / serious adverse device effects (ADE / SADE) reporting using CTCAE/MedDRA coding terms
Safety endpoints of special interest assessment | 16 weeks
  Incidence of tumor lysis syndrome and systemic inflammatory response syndrome.
Clinical endpoint - overall survival | 16 weeks
  A series of secondary efficacy outcome measures will be evaluated based on overall survival from the date of the firststudy treatment and changes in objective response using RECIST (1.1) or iRECIST criteria. The assessed parameterswill be:Overall Survival (OS). Overall survival ( OS ) is defined as the time from randomization to death from any cause, is adirect measure of clinical benefit to a patient.
Clinical endpoint - progression free survival | 16 weeks
  A series of secondary efficacy outcome measures will be evaluated based on overall survival from the date of the firststudy treatment and changes in objective response using RECIST (1.1) or iRECIST criteria. The assessed parameterswill be:Progression Free Survival (PFS) Progression-free survival ( pfs ) is defined as time from randomization until firstevidence of tumour progression or until death from any cause, whichever comes first.
Clinical endpoint - disease control rate | 16 weeks
  A series of secondary efficacy outcome measures will be evaluated based on overall survival from the date of the firststudy treatment and changes in objective response using RECIST (1.1) or iRECIST criteria. The assessed parameterswill be:Disease Control Rate (DCR) Overall response rate (ORR) is defined as the proportion of patients who have a partialor complete response to therapy; it does not include stable disease and is a direct measure of drug tumoricidal activity.In contrast, disease control rate is a composite of ORR and stable disease and is useful to measure the efficacy oftherapies that have tumoristatic effects rather than tumoricidal effects.

SECONDARY OUTCOMES:
Nutritional status | 16 weeks
  Nutritional status will be assessed with PG-SGA scale and via laboratory assessments of changes in serum albumin and CRP concentration. The Scored Patient-Generated Subjective Global Assessment (PG-SGA©) scale will be used. The Scored PG-SGA©includes the four patient-generated historical components (Weight History, Food Intake, Symptoms and Activities andFunction - also known as the PG-SGA Short Form©), the professional part (Diagnosis, Age, Metabolic stress, andPhysical Exam), the Global Assessment (A = well nourished, B = moderately malnourished or suspected malnutrition,C = severely malnourished) and the total numerical score
Patient functioninig with Eastern Cooperative Oncology Group (ECOG) | 16 weeks
  Eastern Cooperative Oncology Group (ECOG) scale describes patient's functioning in terms of ability to care forthemselves, daily activity, and physical ability (walking, working). The scale grades 0 to 5 (0=fully active while 5=dead).
Quality-of-life (QoL) Assessment with EQ-5D-5L scale | 16 weeks
  EQ-5D-5L scale to assess: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimensionhas 5 levels:from no problems to extreme problems.
Quality-of-life (QoL) Assessment with EORTC-QLQ-C30 scale | 16 weeks
  EORTC-QLQ-C30 scale measures cancer patients' physical, psychological and social functions. The EORTC QLQ-C30 comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, fivefunctioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. All of the scales and single-item measures range in score from 0 to 100.Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better stateof the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. aworse state of the patient).
Quality-of-life (QoL) Assessment with EORTC: QLQ-BR23 | 16 weeks
  EORTC: QLQ-BR23 (breast) measuring the quality of life in patients with breast cancer. Each dimension in the scale has four response levels from not at all (1) to very much (4).
Physical performance status assessment with 6 minute walk test (6MWT) | 16 weeks
  The physical performance assessment will be measured with 6-minute walk test (6MWT). 6MWT meassures the distance patient covers when walking in a regular pace in standardized condition. The longerdistance is expected in patients who improve while the poor patient performance and capability, the shorter distancewill be measured.
Muscle performance assessment with a hand grip test | 16 weeks
  The muscle performance assessment will be measured hand grip test. The purpose of this test is to measurethe maximum isometric strength of the hand and forearm muscles. The participant will be asked to squeeze thedynamometer as hard as possible with each of his or her hands in a standing position. The subject squeezes thedynamometer with maximum isometric effort, which is maintained for about 5 seconds. Results for left and right handseparately are recorded in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Ostrowski, MD, Study Director — Immunicom Inc
Locations (5):
- Poland (4):
  - Katedra i Klinika Onkologii UJ CM, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne INTERCOR Sp. z o.o., Bydgoszcz
  - Klinika Pneumonologii, Onkologii i Alergologii SPSK Nr 4 w Lublinie, Lublin
  - Centrum Medyczne Pratia Poznań, Skórzewo
- Altunizade Acıbadem Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No